CLINICAL TRIAL: NCT07360275
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of VCT220 in Participants With Hypertension and Obesity or Overweight.
Brief Title: A Study of VCT220 in Participants With Hypertension and Obesity or Overweight
Acronym: VICTOR-HTN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCT220-II-03
Record Dates: First submitted 2026-01-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VCT220 80mg (Experimental): Participants will receive VCT220 orally everyday. Starting from 20mg and maintaining at 80mg
  Interventions: Drug: VCT220 Tablet
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: VCT220 Placebo Tablet
- VCT220 160mg (1) (Experimental): Participants will receive VCT220 orally everyday. Starting from 20mg and maintaining at 160mg
  Interventions: Drug: VCT220 Tablet
- VCT220 160mg (2) (Experimental): Participants will receive VCT220 orally everyday. Starting from 40mg and maintaining at 160mg
  Interventions: Drug: VCT220 Tablet

INTERVENTIONS:
Drug: VCT220 Tablet — Administered orally, with or without food.
  Arms: VCT220 160mg (1); VCT220 160mg (2); VCT220 80mg
Drug: VCT220 Placebo Tablet — Administered orally, with or without food.
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the safety and efficacy of VCT220 for the treatment of hypertension in participants with obesity or overweight.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants aged 18 to 75 years (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 24 kg/m² at screening.
3. Diagnosed with primary hypertension, with office seated systolic blood pressure (SBP) ≥ 140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg at both screening and baseline.
4. Either treatment-naïve to antihypertensive therapy for ≥ 30 days prior to screening, or receiving a stable dose for ≥ 30 days of one or two of the following classes of antihypertensive medications: renin-angiotensin system inhibitors (ARB/ACEI), calcium channel blockers (CCB), or diuretics.
5. Has at least one self-reported history of unsuccessful weight loss through dietary control.
6. Willing and able to maintain a stable residence and remain contactable throughout the study, and to adhere to regular lifestyle routines as well as dietary and exercise management during the trial.
7. Has a full understanding of the study procedures, is able to communicate effectively with the investigator, understands and is willing to comply with all study requirements, and voluntarily provides written informed consent.

Exclusion Criteria

1. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2).
2. History of or current secondary hypertension.
3. Office seated systolic blood pressure (SBP) ≥ 170 mmHg and/or diastolic blood pressure (DBP) ≥ 110 mmHg at screening or baseline, or presence of a hypertensive emergency.
4. A decrease in office seated SBP of ≥ 20 mmHg or a decrease in office seated DBP of ≥ 10 mmHg at baseline compared with screening.
5. Presence of orthostatic hypotension at screening, defined as a decrease in office SBP of ≥ 15 mmHg or DBP of ≥ 7 mmHg upon transition from the seated to standing position.
6. A difference of ≥ 20 mmHg in office seated SBP between the left and right upper arms at screening or baseline.
7. Treatment with any marketed or investigational drug with a glucagon-like peptide-1 (GLP-1) receptor agonist mechanism within 1 year prior to screening.
8. Self-reported or documented body weight change of ≥ 5 kg within 3 months prior to screening.
9. History of or current type 1 or type 2 diabetes mellitus.
10. History of or current malignancy within the past 5 years, except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
11. History of or current major cardiovascular or cerebrovascular disease.
12. History of or current severe gastrointestinal disease or prior major gastrointestinal surgery.
13. Clinically significant active or unstable severe major depressive disorder or other severe psychiatric disorders within 2 years prior to screening; or any history of suicide attempt.
14. Patient Health Questionnaire-9 (PHQ-9) score ≥ 15 at screening, or a positive response to Item 9.
15. Pregnant or breastfeeding women; or men or women of childbearing potential who are unwilling to use highly effective contraception throughout the study and for 3 months after the last dose, or who plan to conceive, donate sperm, or donate oocytes during this period; or women with a positive pregnancy test at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in office seated systolic blood pressure (SBP) at Week 20 | From baseline to week 20
  Measured In mmHg

SECONDARY OUTCOMES:
Change from baseline in office seated diastolic blood pressure (DBP) at Week 20 | From baseline to week 20
  Measured in mmHg
Change from baseline in 24-hour ambulatory blood pressure monitoring (ABPM) systolic blood pressure and diastolic blood pressure at Week 20 | From baseline to week 20
  Measured in mmHg
Proportion of participants achieving the standard blood pressure target (< 140/90 mmHg) based on office seated blood pressure at Week 20 | From baseline to week 20
  Measured in percentage
Proportion of participants achieving the intensive blood pressure target (< 130/80 mmHg) based on office seated blood pressure at Week 20 | From baseline to week 20
  Measured in percentage
Changes in body weight at week 20 | From baseline to week 20
  Measured in Kg
Adverse events, including treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) | From baseline to week 20
  Count of events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality